CLINICAL TRIAL: NCT01017900
Title: Comparison Between Surgical Excision and Manual Rupture for Dorsal Carpal Ganglion
Brief Title: Surgery Versus Manual Rupture for Dorsal Carpal Ganglion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51-041-11-4-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-23 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Dorsal Carpal Ganglion
Keywords: surgery; manual rupture; dorsal carpal ganglion
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: local excision — surgical excision by orthopaedic surgeon under local anesthesia

SUMMARY:
This study objectives are to compare the efficacy and safety between surgical excision and manual rupture for dorsal carpal ganglion.The participants with dorsal carpal ganglion will be randomized into 2 groups:surgical excision or manual rupture.The patients will be follow-up for at least 1 yr.Telephone interview will be used for outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients with dorsal carpal ganglion

Exclusion Criteria:

* underlying rheumatic condition
* bleeding tendency

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 1,2 and 3 years

SECONDARY OUTCOMES:
time to recurrence | 1,2 and 3 years
DASH score | 1,2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D., Principal Investigator — Department of Orthopaedic Surgery,Faculty of Medicine, Prince of Songkla University, Hat Yai,Songkhla, Thailand 90110
Locations (1):
- Songklanakarind hospital, Hat Yai, Changwat Songkhla, Thailand